CLINICAL TRIAL: NCT05703256
Title: Confirmatory Efficacy Randomized Clinical Trial of Amygdala Neurofeedback for Major Depressive Disorder
Brief Title: Amygdala Neurofeedback for Depression - Large Scale Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kymberly Young (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Kymberly Young, Associate Professor of Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY23010004; R01MH130337 (NIH)
Record Dates: First submitted 2023-01-18; First posted 2023-01-30 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
Keywords: neurofeedback; amygdala; depression; major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive amygdala neurofeedback or yoked sham neurofeedback (seeing the amygdala activity of another participant)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Amygdala real-time fMRI neurofeedback (Experimental): Amygdala neurofeedback - attempt to upregulate the left amygdala during positive autobiographical memory recall via real time fMRI neurofeedback from the amygdala. Two sessions will be performed one week apart.
  Interventions: Device: Amygdala real-time fMRI neurofeedback
- Sham feedback (Sham Comparator): Yoked sham - participants will see the amygdala activity of another subject who completed the intervention. Two sessions will be performed one week apart.
  Interventions: Device: Sham feedback

INTERVENTIONS:
Device: Amygdala real-time fMRI neurofeedback — Participants are shown activity from their left amygdala in real time and are instructed to increase the level of activity in that region by thinking of positive autobiographical memories
  Arms: Amygdala real-time fMRI neurofeedback
Device: Sham feedback — Participants are shown activity from another participant's left amygdala who previously completed the task and are instructed to increase the level of activity in that region by thinking of positive autobiographical memories
  Arms: Sham feedback

SUMMARY:
The goal of this study is to evaluate whether rtfMRI-nf training to increase the amygdala response to positive memories may serve as a stand-alone intervention for major depressive disorder

DETAILED DESCRIPTION:
Previous research has shown that real-time fMRI neurofeedback (rtfMRI-nf) training aimed at increasing the amygdala's response to positive autobiographical memory recall holds therapeutic potential for treating patients with major depressive disorder (MDD), as clinically significant decreases in clinician administered and self-report measures of depression severity were observed following two rtfMRI amygdala neurofeedback sessions. Furthermore, rtfMRI amygdala neurofeedback changed emotional processing towards a positive bias. The goal of the current study is to confirm the clinical efficacy of this intervention in a new sample of depressed participants. Thus, over the course of four years, we will conduct a randomized double-blind clinical trial examining the clinical and cognitive effects of amygdala rtfMRI-nf compared to yoked sham rtfMRI-nf (seeing the amygdala activity of another participant during training) in 200 participants with MDD from the Pittsburgh metropolitan area. Participants will undergo two rtfMRI-nf sessions. Half of the participants will receive amygdala neurofeedback and half will receive yoked sham neurofeedback. Participants will complete the BDI-II monthly for one year following completion of the neurofeedback intervention. The rationale for the proposed research is to provide new insights into possible mechanistic solutions for MDD, and to further guide development of this rtfMRI-nf intervention into a treatment for MDD.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 - 55
* primary diagnosis of MDD and are currently depressed
* able to give written informed consent prior to participation
* unmedicated OR are stable on an antidepressant regime (at least 4 weeks to ensure symptoms are stable). Effective medications will not be discontinued for the purposes of the study.

Exclusion Criteria:

* clinically significant or unstable cardiovascular, pulmonary, endocrine, neurological, gastrointestinal illness or unstable medical disorder
* Current severe DSM-V alcohol or substance use disorder, with the exception of nicotine or caffeine. Clinician will access subjects' alcohol and substance use on a case-by-case to determine whether specific cases of mild or moderate alcohol or substance use would also interfere with the effects of the intervention.
* history of traumatic brain injury
* unable to complete MRI scan due to claustrophobia or general MRI exclusions (e.g., shrapnel inside body)
* currently pregnant or breast feeding
* unable to complete questionnaires written in English
* current (within 3 weeks of testing) use of any antipsychotics, anticonvulsants, stimulants, benzodiazepines, beta-blockers, or other medications (except antidepressants) likely to influence cerebral blood flow. Effective medications will not be discontinued for the purposes of the study.
* diagnosis of psychotic or organic mental disorder, bipolar I or II disorder.
* eye problems or difficulties in corrected vision.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI-II) | baseline vs up to one year
  measures depressive symptoms. The total score will be used, which ranges from 0-63. A total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe. Lower values represent better outcomes.

SECONDARY OUTCOMES:
Life Functioning Questionnaire (LFQ) | baseline vs up to one year
  measures ability to function in daily life. The total score will be used, which ranges from 14-56. A total score of 14-27 indicates no problems, and a score of 28+ indicates some impairment. Lower values represent better outcomes.

OTHER OUTCOMES:
Autobiographical Memory Test | baseline vs one month
  measures memory specificity. Participants are asked to recall a memory in response to 18 cue words. The number of specific memories is determined and reported. Scores can range from 0-18 and higher scores represent better memory performance.

CONTACTS AND LOCATIONS:
Overall Officials: Kymberly Young, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All fMRI, BDI and LFQ scores for IPD will be made available through the NDAR data repository
Time Frame: New data will be uploaded every 6 months and be available indefinitely
Access Criteria: Users with NDA credentials may submit Data Access Requests. Data Access Requests for a given NDA Permission Group are reviewed by an NIH-staffed Data Access Committee.
URL: https://nda.nih.gov

REFERENCES:
- [Background] Young KD, Zotev V, Phillips R, Misaki M, Yuan H, Drevets WC, Bodurka J. Real-time FMRI neurofeedback training of amygdala activity in patients with major depressive disorder. PLoS One. 2014 Feb 11;9(2):e88785. doi: 10.1371/journal.pone.0088785. eCollection 2014. PMID 24523939
- [Background] Young KD, Siegle GJ, Zotev V, Phillips R, Misaki M, Yuan H, Drevets WC, Bodurka J. Randomized Clinical Trial of Real-Time fMRI Amygdala Neurofeedback for Major Depressive Disorder: Effects on Symptoms and Autobiographical Memory Recall. Am J Psychiatry. 2017 Aug 1;174(8):748-755. doi: 10.1176/appi.ajp.2017.16060637. Epub 2017 Apr 14. PMID 28407727
- [Background] Young KD, Misaki M, Harmer CJ, Victor T, Zotev V, Phillips R, Siegle GJ, Drevets WC, Bodurka J. Real-Time Functional Magnetic Resonance Imaging Amygdala Neurofeedback Changes Positive Information Processing in Major Depressive Disorder. Biol Psychiatry. 2017 Oct 15;82(8):578-586. doi: 10.1016/j.biopsych.2017.03.013. Epub 2017 Mar 28. PMID 28476207